CLINICAL TRIAL: NCT02688439
Title: Effect of Leg Positioning and Tourniquet Inflation on Onset and Duration of Ultrasound Guided Sciatic Nerve Block After Injection of Local Anesthetic
Brief Title: Ultrasound Guided Sciatic Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-01327
Record Dates: First submitted 2016-01-20; First posted 2016-02-23 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Sciatic Nerve

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Leg in a neutral position (Active Comparator): Sciatic nerve block, with leg kept in a neutral position after anesthesia (control group)
  Interventions: Other: Sciatic Nerve block; Other: Leg in a neutral position
- Leg raised 30° (Experimental): Sciatic nerve block, with leg raised 30° by placing the back of the foot over a support placed on the OR table and maintained in that position for 15 min
  Interventions: Other: Sciatic Nerve block; Other: Leg raised 30°
- Distal tourniquet placed on the lower part of the leg (Experimental): Sciatic nerve block, and distal tourniquet placed on the lower part of the leg (upper part of the tourniquet being about 4-6 inches from the ankle) with the leg in a neutral position.
  Interventions: Other: Sciatic Nerve block; Other: Distal tourniquet placed on the lower part of the leg; Other: Leg in a neutral position

INTERVENTIONS:
Other: Sciatic Nerve block
Other: Leg raised 30°
  Arms: Leg raised 30°
Other: Distal tourniquet placed on the lower part of the leg
  Arms: Distal tourniquet placed on the lower part of the leg
Other: Leg in a neutral position
  Arms: Distal tourniquet placed on the lower part of the leg; Leg in a neutral position

SUMMARY:
The primary purpose of this study is to determine whether the leg positioning or distal tourniquet used during the injection of local anesthetic may decrease the onset time and prolong the duration of analgesia of ultrasound-guided Sciatic Nerve Block (SNB) with popliteal approach. Patients will be divided randomly into three groups: group 1 will receive sciatic nerve block, with leg kept in a neutral position after anesthesia (control group); group 2 will receive the same anesthesia, with leg raised 30° by placing the back of the foot over a support placed on the OR table and maintained in that position for 15 min; and patients in group 3 will receive the same anesthesia, and distal tourniquet placed on the lower part of the leg (upper part of the tourniquet being about 4-6 inches from the ankle) with the leg in a neutral position

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective foot surgery under ultrasound guided popliteal sciatic/saphenous block
* American Society of Anesthesiologist physical status 1-3, meaning patients who are either completely or their systemic disease(s), if they have is (are) under control with medications or other means.
* Have capacity to provide informed consent.

Exclusion Criteria:

* clinically significant coagulopathy (impaired blood clotting)
* infection at injection site
* allergy to local anesthetics
* severe cardiopulmonary disease (heart and lung disease)
* body mass index >35 kg.m2
* known neuropathies (degenerative, infectious and traumatic peripheral nerve diseases)
* who are receiving opioids for chronic analgesic therapy at the time of contemplated surgery
* Patients with history of AIDS, tuberculosis, and other infections
* active and/or unstable cardiac, renal, pulmonary and neurologic disorders will be excluded from the study. This includes patients in heart failure having limited exercise ability, end stage renal failure on dialysis treatment, recent stroke etc.
* Vulnerable subjects (children, pregnant subjects, prisoners, mentally impaired) also will not be included in the study.
* Subjects who do not understand or speak English

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-03; Primary Completion 2017-12-29 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of Sensory block by measuring decrease in sensation on the scale of 0 to 5 (0 being no sensation; 5 being most sensation) as compared to the other foot. | 15 Minutes
Evaluation of motor block evaluated by measuring movement on the scale of 0 to 5 as compared to the other foot. | 15 Minutes
Level of pain measured on a scale of 0 to 10 (0 being no pain; 10 being most pain) prior to first pain killer | 15 Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Levon Capan, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States